CLINICAL TRIAL: NCT03530553
Title: Using the Hunt Motivational Scale to Aid in Weight Loss and Weight Maintenance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Penn Medicine Princeton Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN 2337
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: There are two arms in this study. One group will receive the HMS and the other will not and will receive standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): The treatment arm will receive the HMS as well as standard of care of the weight management program.
  Interventions: Other: Hunt Motivational Scale
- Control arm (No Intervention): The control arm will not receive the HMS and will receive standard of care.

INTERVENTIONS:
Other: Hunt Motivational Scale — The Hunt Motivational Scale is a tool to help facilitate weight loss and motivate patients to track, plan, and practice healthy weight loss and weight maintenance practices.
  Arms: Treatment arm

SUMMARY:
In this study, we plan to determine the efficacy of the Hunt Motivational Scale as a tool for weight loss compared to standard of care in the Penn Medicine Princeton Health weight management program.

DETAILED DESCRIPTION:
Obesity is rising at alarming rates, currently at nearly 40%. There are very few tools, specifically questionnaires, for healthcare providers to help their patients lose weight or maintain their weight loss. The Hunt Motivational Scale is one such tool to help patients identify areas that need improvement in order to aid in weight loss and weight maintenance. The HMS is designed to motivate patients to track, plan, and practice other healthy weight loss and weight maintenance practices so that they will have success.

In this study, approximately 75 subjects in the Penn Medicine Princeton Health weight management program will be randomly assigned to either receive the HMS or not (standard of care). They will be followed for a period of six months at the end of which it will be determined whether the group that received the HMS lost more weight than the control group.

ELIGIBILITY:
Inclusion Criteria:

* patient in weight management program at Penn Medicine Princeton Health

Exclusion Criteria:

* does not have a visit every three to four weeks
* not in active weight loss phase of the program
* diminished intellectual capacity to complete questionnaire i.e. Down's syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-10-11 (Estimated); Study Completion 2018-10-11 (Estimated)

PRIMARY OUTCOMES:
Weight loss | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine Princeton Health, Plainsboro, New Jersey, United States